CLINICAL TRIAL: NCT00163150
Title: Lacunar-Brain Infarction Cerebral Hyperactivity And Atorvastatin Trial. A Placebo-Controlled Trial Of High-Dose Atorvastatin In Patients With Cerebral Small Vessel Disease.
Brief Title: Vasomotor Reactivity In Cerebral Small Vessel Disease And New Approach To Treat Lacunar Stroke
Acronym: LA BICHAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581063
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cerebrovascular Accident; Hypercholesterolemia
MeSH Terms: conditions — Stroke; Hypercholesterolemia | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
The main purpose of this study is to evaluate the efficacy of atorvastatin treatment during 3 months (80mg/day) on cerebral vasoreactivity (CVR) in lacunar patients.

ELIGIBILITY:
Inclusion Criteria:

* clinically defined lacunar syndrome 3 months before inclusion
* small deep infarct on diffusion MRI (Diffusion Weighted Imaging)
* no atherothrombotic, cardio-embolic, or other rarer cause.

Exclusion Criteria:

* patients with past coronary event
* contra-indication for assessment of vasomotor reactivity
* patients being on statin therapy at the time of brain infarction
* contra-indication for statin therapy
* patient still under statin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128
Dates: Start 2003-06; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of atorvastatin treatment during 3 months (80mg/day) on cerebral vasoreactivity (CVR) in lacunar patients. CVR, humeral and carotid vasoreactivity will be measured in all patients at M0 and M3.

SECONDARY OUTCOMES:
Evaluate the efficacy of atorvastatin treatment during 3 months (80mg/day) on endothelium dependant and independent vasomotoricity of humeral and / or common carotid artery (according to validation study) in lacunar patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

REFERENCES:
- [Derived] Lavallee PC, Labreuche J, Gongora-Rivera F, Jaramillo A, Brenner D, Klein IF, Touboul PJ, Vicaut E, Amarenco P; Lacunar-BICHAT Investigators. Placebo-controlled trial of high-dose atorvastatin in patients with severe cerebral small vessel disease. Stroke. 2009 May;40(5):1721-8. doi: 10.1161/STROKEAHA.108.540088. Epub 2009 Mar 12. PMID 19286582
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581063&StudyName=Vasomotor+Reactivity+In+Cerebral+Small+Vessel+Disease+And+New+Approach+To+Treat+Lacunar+Stroke+